CLINICAL TRIAL: NCT01195285
Title: Single-Incision Laparoscopic Cholecystectomy Versus Traditional Laparoscopic Cholecystectomy: A Randomized Prospective Trial
Brief Title: Single-Incision Laparoscopic Cholecystectomy Versus Traditional Laparoscopic Cholecystectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decisions based on slow enrollment.
Sponsor: Saint Luke's Health System (Other)
Collaborators: Tyco Healthcare Group LP (d/b/a Covidien) (Unknown)
Responsible Party: Kimberly Brown, MD, Saint Luke's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-423
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2011-08

CONDITIONS: Biliary Dyskinesia; Gallstones; Cholecystitis; Cholelithiasis
Keywords: Laparoscopic cholecystectomy; Quality of life; Biliary Cholic; Chronic Cholecystitis; Symptomatic Cholelithiasis
MeSH Terms: conditions — Biliary Dyskinesia; Gallstones; Cholecystitis; Cholelithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-Incision Laparoscopic Cholecsytectomy (SILS) (Active Comparator)
  Interventions: Procedure: Single-Incision Laparoscopic Surgery cholecystectomy
- Traditional Laparoscopic Cholecystectomy (TLC) (Active Comparator)
  Interventions: Procedure: Traditional Laparoscopic Cholecystectomy (TLC)

INTERVENTIONS:
Procedure: Single-Incision Laparoscopic Surgery cholecystectomy — Laparoscopic Cholecystectomy
  Arms: Single-Incision Laparoscopic Cholecsytectomy (SILS)
Procedure: Traditional Laparoscopic Cholecystectomy (TLC) — Laparoscopic Cholecystectomy
  Arms: Traditional Laparoscopic Cholecystectomy (TLC)

SUMMARY:
This study will compare Single Incision Laparoscopic Surgery (SILS) cholecystectomy to traditional laparoscopic cholecystectomy (LC), focusing on patient-reported outcomes and cost.

DETAILED DESCRIPTION:
Single-Incision Laparoscopic Surgery (SILS) is accepted as a form of surgical treatment. Traditional laparoscopic cholecystectomy (TLC) is well tolerated, with a low complication risk and high patient satisfaction; thus a SILS procedure needs to be at least equivalent to be a justifiable replacement, and should not result in higher costs.

ELIGIBILITY:
Inclusion Criteria:

* Patient recommended to undergo cholecystectomy
* Patient age 18-80
* Patient competent to give his/her own informed consent
* Patient speaks English without the need for an interpreter

Exclusion Criteria:

* Additional procedures planned during same surgery
* Patient deemed inappropriate for TLC or SILS cholecystectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cost associated with performance of the procedure and post-operative care until discharge | 4 weeks

SECONDARY OUTCOMES:
Pain scale reported by patient at discharge, 24 and 48 hours | 24 hours and 48 hours
Amount of pain medicine required during 48 hours after surgery | 48 hours
Major and minor gastrointestinal surgical complications, including conversion | 4 weeks
Quality of Life | 2 weeks and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly M Brown, BS, MD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

REFERENCES:
- [Background] Single-incision Laparoscopic Surgery Launched at St. Louis University Hospital. www.news-medical.net. April, 2009
- [Background] Chamberlain RS, Sakpal SV. A comprehensive review of single-incision laparoscopic surgery (SILS) and natural orifice transluminal endoscopic surgery (NOTES) techniques for cholecystectomy. J Gastrointest Surg. 2009 Sep;13(9):1733-40. doi: 10.1007/s11605-009-0902-y. Epub 2009 May 2. PMID 19412642
- [Background] Hodgett SE, Hernandez JM, Morton CA, Ross SB, Albrink M, Rosemurgy AS. Laparoendoscopic single site (LESS) cholecystectomy. J Gastrointest Surg. 2009 Feb;13(2):188-92. doi: 10.1007/s11605-008-0735-0. Epub 2008 Nov 22. PMID 19031097